CLINICAL TRIAL: NCT06476769
Title: Combined Effects of Blow Bottle Device and Postural Drainage in Moderate to Severe Elderly COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0376
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Dyspnea; Postural drainage
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Drainage, Postural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blow bottle technique (Experimental): There were 20 patients in group A received blow bottle device and postural drainage for 20- 25 minutes per session twice a day for 4 days per week, for 8 weeks.
  Interventions: Other: blow bottle technique
- percussion (Active Comparator): There were 20 patients in group B received postural drainage with percussion for 20- 25 minutes per session twice a day for 4 days per week, for 8 weeks.
  Interventions: Other: percussion

INTERVENTIONS:
Other: blow bottle technique — There were 20 patients in group A received blow bottle device and postural drainage for 20- 25 minutes per session twice a day for 4 days per week, for 8 weeks.
  Other Names: postural drainage
  Arms: blow bottle technique
Other: percussion — Group B: There were 20 patients in group B received postural drainage with percussion for 20- 25 minutes per session twice a day for 4 days per week, for 8 weeks.
  Other Names: postural drainage
  Arms: percussion

SUMMARY:
It will be a randomized clinical trial. Age of selected subjects will be between 40 to 70 years. Data will be collected from Wazirabad institute of cardiology. There will be 2 groups i.e. group A will receive combination of blow bottle technique and postural drainage and group B will receive postural drainage. Spirometer will be used to evaluate pulmonary functions and breathless, cough and sputum scale (BCSS) will be used to evaluate the improvement in sputum diary of patients. Interventions will be given to the patients for 20-25 minutes twice a day for 6 days per week. After data collection, data will be analyzed using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed moderate to severe GOLD (2017) COPD
* 40-60 years old
* Both male and female
* Patients hemodynamically stable
* PFT showing irreversible airflow limitation.

Exclusion Criteria:

* Type II diabetic mellitus
* Systemic illness
* Thoracic deformation or rib fracture.
* Pulmonale decompensation and signs of an unstable heart condition.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Breathlessness cough sputum scale | 4 weeks
  Breathlessness, Cough and Sputum scale (BCSS) was developed to effectively measure the severity of respiratory symptoms. The BCSS records symptoms in a 5-point Likert like scale in which zero represents improvement symptoms and scores towards 4 indicating worsening of symptoms. It is commonly used in patients with COPD. BCSS provides a simple and robust quantification of symptoms that is sensitive to the effects of treatment and could therefore be used to assess therapeutic interventions. It has good reliability and validity for use in patients with respiratory disorders.
Modified borg RPE scale: | 4 weeks
  The Modified Borg Dyspnea Scale (MBS) is rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise, one of the most common and frequently used measures to assess the severity of dyspnea.
Incentive spirometry | 4 weeks
  Incentive spirometry is frequently used after thoracic surgery as an adjunct to physiotherapy. Despite its widespread use, it has remained challenging to demonstrate a clinical benefit in terms of either incidence of pulmonary complications or hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Wazirabad Institute of Cardiology, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kullowatz A, Kanniess F, Dahme B, Magnussen H, Ritz T. Association of depression and anxiety with health care use and quality of life in asthma patients. Respir Med. 2007 Mar;101(3):638-44. doi: 10.1016/j.rmed.2006.06.002. Epub 2006 Aug 7. PMID 16891108
- [Background] Goodwin RD, Eaton WW. Asthma and the risk of panic attacks among adults in the community. Psychol Med. 2003 Jul;33(5):879-85. doi: 10.1017/s0033291703007633. PMID 12877402
- [Background] Wright RJ, Rodriguez M, Cohen S. Review of psychosocial stress and asthma: an integrated biopsychosocial approach. Thorax. 1998 Dec;53(12):1066-74. doi: 10.1136/thx.53.12.1066. PMID 10195081